CLINICAL TRIAL: NCT04242056
Title: To Study the Pathophysiological Features of Multiple Sclerosis: Combined Multi-modalities of Amyloid and Tau Images Associated With Serum Neurofilament Light Chain Levels
Brief Title: To Study the Pathophysiological Features of Multiple Sclerosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsu, Jung-Lung, MD, Associate Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201802146A0
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis; Neurofilament Light Chain; Glial Fibrillary Acidic Protein
MeSH Terms: conditions — Multiple Sclerosis; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Using image to diagnosis Multiple sclerosis (MS) (Other): In current study, we will enroll 38 patients with MS and evaluate their clinical severity; measure the WM lesion and disease activity by magnetic resonance imaging (MRI); myelination state and amyloid deposition by amyloid PET scan; tau deposition by state of-art tau PET scan
  Interventions: Drug: 18F-PM-PBB3

INTERVENTIONS:
Drug: 18F-PM-PBB3 — 18F-PM-PBB3 brain PET studies will be conducted for 38 subjects. Dynamic PET/MRI studies will be collected by PET/MRI scanner for 100 minutes (4×15 s, 8×30 s, 960 s, 2×180 s, 8300 s, 3×600 s). Volumes of interest (VOIs) will be delineated from corresponding MR images by manual including bilateral frontal, parietal, mesial temporal, lateral temporal, hippocampal, occipital, anterior cingulate, posterior cingulate, cerebellum areas, and genu region of white matter. The DVRs will be computed from Logan graphic analysis by using cerebellum as reference input.
  SUVR of every cortical VOI to the gray matter of cerebellum will be calculated from nine 10-min dynamic image sets.

SUMMARY:
Multiple sclerosis (MS) is the most common chronic inflammatory disease of the central nervous system1, whose demyelination is the pathological hallmark. MS is characterized by neuroinflammation, demyelination, axonal damage, and neurodegeneration2. The demyelination state in brain and the clinical course are difficult to predict in the early stage of disease. Recently, several neuroimaging and fluid biomarkers had been explored in MS. Using brain amyloid positron emission tomography (PET) in active MS had showed that both the damage sites and normal appearance white matter had a lower intensity than non-active MS. The result suggests a predictive role that the intensity from amyloid PET could reflect the disease activity and link to early myelin damage. The levels of tau protein in cerebrospinal fluid (CSF) had also been showed a negative correlation with brain atrophy, which is a prognostic marker for MS. In fluid biomarkers, both neurofilament light chain (NfL) and glial fibrillary acidic protein (GFAP) had been used in MS and reported correlations with disease severity, the extent of neuroinflammation and progression. In current study, investigator will enroll 38 participants with MS and evaluate their clinical severity; measure the WM lesion and disease activity by magnetic resonance imaging (MRI); myelination state and amyloid deposition by amyloid PET scan; tau deposition by state of-art tau PET scan. Investigator also measure the serum levels of NfL and GFAP as the index of axonal injury and disease activity. The relationship between disease severity, brain myelination, tau deposition and serum levels of NfL will be discuss.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-75 years old
2. Multiple Sclerosis patients

Exclusion Criteria:

1. Implantation of metal devices including cardiac pacemaker, intravascular metal devices.
2. Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes, acute myocardial infarction, poorly controlled diabetes, previous severe head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases.
3. Major psychiatric disorders, drug or alcohol abuse and major depression
4. Pregnant women or breast- feeding women.
5. Patients in whom MRI was contraindicated or patient had claustrophobia.
6. History of severe allergic or anaphylactic reactions particularly to the tested drugs.
7. History of positive test for human immunodeficiency virus (HIV).
8. Indication of impaired liver function as shown by an abnormal liver function profile at screening (eg. repeated values of aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≧ 3X the upper limit of normal values).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between hyperintensity lesions in FLAIR MRI and demyelination in amyloid PET image | 3 years
  Investigator would be able to find the topographical correlation between hyperintensity lesions in FLAIR MRI and hypointensity lesions in amyloid PET, measurement by overlapping volume (ml) and overlapping ratio (%)

SECONDARY OUTCOMES:
Correlation between clinical parameters (EDSS) and hyperintensity lesions in FLAIR MRI and hyperintensity region of tau PET image light chain and GFAP levels. | 3 years
  Investigator would be able to find the EDSS correlation between whole brain hyperintensity lesions in FLAIR MRI (ml) and hyperintensity regions of tau PETwe will take this advantage to perform the study and explore the relationship between serum neruofilament light chain and GFAP levels.
Correlation between clinical parameters (EDSS) and serum NfL levels | 3 years
  Investigator would be able to find the EDSS correlation between EDSS and serum NfL levels